CLINICAL TRIAL: NCT04520204
Title: Russian Registry of Acute Myocardial Infarction
Brief Title: National, Multi-center, Prospective, and Retrospective Cohort Study.
Acronym: REGION
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Healthy Future (Other)
Responsible Party: Sponsor
Other Study IDs: AMI 05.2020
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
National, multi-center, observational, prospective, and retrospective cohort study. The study does not provide for intervention in routine clinical practice.

Key goals:

• Obtaining real-world evidence on the diagnosis and treatment of AIM in Russian hospitals, including both long- and short-term findings and outcomes (i.e. during hospitalization,

and 6-12 months after the diagnosis establishment).

* Evaluation of the applied approaches to the management of AIM patients for compliance with the clinical recommendations across various hospitals, with a breakdown by equipment status;
* Assessment of patients' treatment adherence after 6 and 12 months.

The expected project duration is 3 years. The study subjects will be recruited during the first 24 months unless the investigators decide to terminate or extend the study period. The period of observation for each patient is 6 to 12 months. The project involves retrospective and prospective collection of information from medical records. All patient data shall be recorded by the Investigator into an approved electronic case report form (eCRF).

Recruitment period: 2020-2022. Expected number of subjects: 10,000.

DETAILED DESCRIPTION:
The Russian Registry of Acute Myocardial Infarction study is an independent study initiated by the investigators;

The partner inpatient hospitals will provide data on every patient with known acute myocardial infarction (I21) admitted between days 1 and 10 of each month during the recruitment period.The Russian Registry of Acute Myocardial Infarction study is an independent study initiated by the investigators;

For every engaged hospital (medical center) the investigators will designate a 2-3 person task team, including a Team Leader;

The participants shall be kept informed and coordinated via email and messengers. The website of the Russian Society of Emergency Cardiology.

The study will be hosted by the CRM Quinta® platform.

Administration, data entry monitoring, and statistical processing will be carried out by Aston Consulting (a certified personal data operator.)

AO Aston Consulting has a license for storage and processing of personal data in accordance with the applicable legislation.

PATIENTS.

INCLUSION CRITERIA

1. Diagnosed acute ST-elevation myocardial infarction (STEMI) or non-ST elevation myocardial infarction (NSTEMI) (ICD 10 I21 ); the diagnosis is established based on the Fourth Universal Definition of Myocardial Infarction Guidelines 2018 .

EXCLUSION CRITERIA

1. A patient or his/her legal representative did not sign IC.

STUDY ASSESSMENTS

The following information will be collected and entered into CRF: Full name

Residential address

Phone number of patients or their legal representatives' Demographic profile. Weight, height

Social status (education, job title, occupation status)

Co-morbidities

Clinical signs and symptoms

Drug therapy.

Clinical outcomes during the hospital stay.

Drug therapy and clinical outcomes in 6 and 12 months after the diagnosis establishment.

Hospitals wishing to join the study must contact any of the project coordinators and complete the Participation questionnaire (Appendix 4).

The Registry enrolment process starts in 2020 and will continue for 24 months. The hospitals that will not be able to start the enrolment in 2020 will have the chance to do it before December 31, 2022, and perform the follow-up monitoring for the next 12 months.

At the moment of the enrolment, the patient's data are to be entered into the online database. Any new data that might appear during the hospital stay will be successively or immediately entered into the database at the moment of the patient's death/discharge. The data received during an in-person or a phone contact 6 or 12 months after the enrolment will also be entered into the database.

Shall the initiators have any questions regarding the entered data, they will ask the participants to elaborate, clarify, or correct the data.

If the patient dies before the enrolment to the study, his/her data shall be entered into the database retrospectively.

The patients (or their legal representatives) enrolled to the Registry must be kept informed about the inclusion in this observational program and give their written consent for participation (patients who died or are otherwise unable to sign the consent to the processing of personal data will be enrolled on a de-identified basis.)

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosed acute ST-elevation myocardial infarction (STEMI) or non-ST elevation myocardial infarction (NSTEMI) (ICD 10 I21); the diagnosis is established based on the Fourth Universal Definition of Myocardial Infarction Guidelines 2018 .

The diagnosed patient was admitted to the hospital between days 1 and 10 of the current mont.

Exclusion Criteria:

1. A patient or his/her legal representative did not sign the IC.

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients 18+1. Diagnosed acute ST-elevation myocardial infarction (STEMI) or non-ST elevation myocardial infarction (NSTEMI) (ICD 10 I21); the diagnosis is established based on the Fourth Universal Definition of Myocardial Infarction Guidelines 2018 and signed ( or his/her legal representative) informed consent
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Monitoring of the patient | 12 monthes
  Recording of all events that occur with the patient for 12 months from the moment of diagnosis Acute myocardial infarction : repeated heart attack, change of therapy, complications from the cardiovascular system, death

SECONDARY OUTCOMES:
Frequency of the following episodes 2. The proportion of patients who continue taking statins, antiplatelets, and drugs from other groups 6 months or 1 year post-discharge. | 12 monthes
  Record the f- recurrent MI
  * heart failure
  * ischemic stroke
  * clinically significant bleeding
  * unplanned revascularisation post-discharge frequency of complications:

CONTACTS AND LOCATIONS:
Overall Officials: Pevzner, Principal Investigator — Myasnikov Institute of Clinical Cardiology
Locations (1):
- Federal State Budgetary Institution NATIONAL MEDICAL CENTER CARDIOLOGY RESEARCH CENTER Ministry of Health of the Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No